CLINICAL TRIAL: NCT04172662
Title: Music Therapy as an Adjunct in Cardiac Implantable Electronic Device (CIED) Lead Extraction Procedures
Brief Title: Music Therapy as an Adjunct in CIED Lead Extraction Procedures
Acronym: MATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Academy of Music (Other)
Responsible Party: Principal Investigator, Sigrun Halvorsen, Professor MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/168
Record Dates: First submitted 2019-10-04; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: C.Surgical Procedure; Stress; Pain, Procedural; Anxiety
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy group (Experimental): Receive Music therapy in addition to standard treatment
  Interventions: Behavioral: Facilitated Music Listening
- Control group (No Intervention): Receive standard treatment

INTERVENTIONS:
Behavioral: Facilitated Music Listening — The patient gets a preparatory session with the music therapist one day before the invasive procedure, where individual assessment is made based on a biopsychosocial approach. Sequences of facilitated Music listening is provided during the pre-, peri and postoperative phase, and a closing dialog performed postoperatively. Patient-preferred music is chosen from a limited set of playlists provided on the app The Music Star.
  Other Names: Music therapy
  Arms: Music therapy group

SUMMARY:
The study will investigate possible effects of music therapy as an adjunct in an invasive cardiac procedure where infected or broken pacemaker leads, or leads from implantable cardioverter-defibrillators are removed from inside the heart through the vein. The procedure is performed in local anaesthesia with the patient awake. Analgesic and anxiolytic drugs are given at the start of the procedure, and repeated if needed. In spite of the drugs, most patients will experience som degree of pain and/or anxiety and increased stress during the procedure. The music therapy intervention contains individually facilitated music listening and coping techniques, aiming to regulate stress responses. The music listening and guidance is provided by a certified music therapist before, during and after the invasive procedure.

DETAILED DESCRIPTION:
See study protocol

ELIGIBILITY:
Inclusion Criteria:

1. Planned pacemaker or intracardiac defibrillator (ICD) lead extraction performed in local anaesthesia.
2. Lead implanted > 12 months ago
3. Able to speak and read Norwegian
4. Willing to participate All inclusion criteria must be fulfilled.

Exclusion Criteria:

1. Significant hearing impairment
2. Previous and/or acute psychiatric diagnosis
3. Cognitive and mental deficits or impaired functioning

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with pain management during the procedure | 1 hour after completion of the procedure
  10-point visual numeric scale, previously used in comparable studies. One represented very dissatisfied and 10 very satisfied
Patient experience of pain intensity during the procedure | Mean pain intensity during the procedure
  Numeric Rating Scale (NRS, 0-10)

SECONDARY OUTCOMES:
Patient experience of anxiety level during the procedure | Mean anxiety level during the procedure
  Numeric Rating Scale (NRS, 0-10)
Effect on vital sign | Mean arterial blood pressure during the procedure
  Mean arterial blood pressure during the procedure
Consumption of analgetic drugs during the procedure | Total amount of analgesic drug (fentanyl) given throughout the procedure
  Total need for fentanyl during the procedure, measured in mg

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Halvorsen, Prof. MD PhD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital, Ullevål, Hjertemedisinsk avdeling, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No